CLINICAL TRIAL: NCT03322215
Title: A Phase 2, International, Multicenter, Open-labeled, Randomized Trial of PAlbociclib and Fulvestrant vs. Standard Oral Capecitabine In Patients With Hormone Receptor (HR)+ / HER2- Advanced Breast Cancer and Documented Endocrine Resistance
Brief Title: HR+/HER2- Advanced Breast Cancer and Endocrine Resistance
Acronym: PASIPHAE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Theodoros Foukakis (Other)
Responsible Party: Sponsor-Investigator, Theodoros Foukakis, Principal Investigator, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-002893-11
Record Dates: First submitted 2017-09-28; First posted 2017-10-26 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer Metastatic
Keywords: palbociclib; fulvestrant; capecitabine
MeSH Terms: interventions — palbociclib; Fulvestrant; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Palbociclib and fulvestrant (Experimental): Combination of palbociclib and fulvestrant
  Palbociclib:
  125 mg capsule administered orally once daily for 21 consecutive days followed by 7 days off treatment. Dose modification is recommended based on individual safety and tolerability.
  Fulvestrant:
  500 mg administered intramuscularly on days 1 and 15 of cycle 1, and then on day 1 of each subsequent 28-day cycle.
  Interventions: Drug: Palbociclib; Drug: Fulvestrant
- Capecitabine (Active Comparator): 1,000 mg/m2 tablet administered orally twice daily for 2 weeks followed by one week of rest. Depending on adverse reactions, both dose escalation and dose reductions will be performed.
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Palbociclib — 75-125 mg capsule orally once daily for 21 consecutive Days followed by 7 Days of treatment.
  Other Names: Ibrance
  Arms: Palbociclib and fulvestrant
Drug: Fulvestrant — 500 mg intramuscularly Days 1 and 15 of cycle 1, and then on Day 1 of each subsequent 28-days cycle.
  Other Names: Faslodex
  Arms: Palbociclib and fulvestrant
Drug: Capecitabine — Oral tablet 500 - 1,250 mg/m2 twice Daily, for 2 weeks followed by 1 week of rest.
  Other Names: Xeloda
  Arms: Capecitabine

SUMMARY:
This is a randomized, 2-arm, open-label, multicenter, international phase II trial. A total of 196 patients will be included.

The study will include patients with metastatic Hormone Receptor positive / Human Epidermal Growth Factor Receptor (HER2) negative breast cancer with progressive disease after endocrine treatment.

Patients will be randomized (1:1) between two treatment arms: A. palbociclib + fulvestrant and b. capecitabine.

ELIGIBILITY:
Inclusion Criteria:

1. Women 18 years or older.
2. Postmenopausal, defined by at least one of the following criteria:

   1. Prior bilateral oophorectomy
   2. Age ≥60
   3. Age <60 and amenorrhea for 12 or more months (in the absence of chemotherapy, tamoxifen, toremifene, or ovarian suppression) and FSH and estradiol in the postmenopausal range according to the local laboratory reference. Note: For women with therapy-induced amenorrhea, serial measurements of FSH and/or estradiol are needed to ensure postmenopausal status. OR Pre/perimenopausal if treated with goserelin that was initiated at least 4 weeks prior to randomization.
3. Locally advanced or metastatic breast cancer deemed not amenable to curative surgery or curative radiation therapy.
4. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
5. Known estrogen-receptor positive and/or progesterone receptor positive breast cancer reported by local laboratory.
6. Known HER2-negative breast cancer defined as a negative in situ hybridization test or an IHC status of 0, 1+ or 2+. If IHC is 2+, a negative in situ hybridization (FISH, CISH, or SISH) test is required by local laboratory testing.
7. Documented resistance to endocrine therapy (tamoxifen or aromatase inhibitors) defined as:

   1. Recurrence while on or within 12 months after the end of adjuvant endocrine treatment OR
   2. Progression while on or within 1 month after the end of endocrine treatment for advanced disease
8. Previous chemotherapy for breast cancer including an anthracycline and a taxane (only one line for metastatic disease) is permitted.
9. Radiological or other objective evidence (eg. new skin lesions or new lymph node lesions) of recurrence during or after the most recent systemic therapy for recurrent / metastatic disease prior to randomization.
10. At least one tumor lesion accessible for biopsy that is a non-bone lesion or a predominantly lytic bone lesion, and that measures at least 10 mm in largest diameter. This lesion must not have been treated previously with irradiation (although the area may have been irradiated before the occurrence of the lesion).
11. Patient is interested to participate in the trial, including the obligatory biopsies at a metastatic site/site before the start of study treatment.
12. Clinically and/or radiographically documented measurable disease according to RECIST v1.1 criteria or bone-only disease with at least one predominantly lytic or mixed bone lesion. For measurable disease, at least one site of disease must have largest tumor diameter of at least:

    1. 10 mm if measured by CT-scan, ultrasound, or physical exam
    2. 20 mm if measured by Chest X-ray
    3. 15 mm if suspiciously enlarged lymph node (short axis) see Eisenhauer et al. for more details All radiology studies must be performed within 28 days prior to registration (35 days if negative).
13. Adequate bone-marrow, hepatic and renal function defined as laboratory tests within 7 days prior to enrollment:

    1. Hematology: Absolute granulocytes > 1.5 x 109/L, Platelets > 100 x 109/L
    2. Biochemistry: Bilirubin ≤ 1.5 x upper limit of normal (ULN), Serum creatinine ≤ 1.5 x ULN.
14. 14. APTT and INR ≤ 1.5 x ULN or institution accepted values for biopsy within 7 days prior to enrollment.
15. Signed written informed consent provided by the patient.

Exclusion Criteria:

1. Previous treatment with a CDK4/6 inhibitor, mTOR or PI3K inhibitor, fulvestrant or capecitabine. Short-term (<28 days) exposure to mTOR or PI3K inhibitor in the (neo)adjuvant setting is allowed.
2. More than one prior chemotherapy lines for metastatic breast cancer. Previous (neo)adjuvant chemotherapy or for radically treated local or regional relapse is allowed in addition to one prior chemotherapy line for metastatic breast cancer Note: A chemotherapy line in advanced disease is an anticancer regimen that contains at least one chemotherapy agent and is given for 21 days or longer. If a cytotoxic chemotherapy regimen was discontinued for a reason other than disease progression and the decision for its discontinuation was taken within 21 days after starting it, then this regimen does not count as a "prior line of chemotherapy". Chemotherapy regimens composed of more than one drug are considered as one line of therapy.
3. No measurable lesions amenable to biopsy (e.g. pleural effusion, ascites, skin rash, sclerotic bone etc).
4. CNS metastases unless asymptomatic and adequately controlled with surgery or radiotherapy. Stable CNS disease is defined as CNS metastases or cord compression that have been definitively treated and the patient is clinically stable off anticonvulsants and steroids for at least 4 weeks before randomization.
5. Leptomeningeal carcinomatosis
6. Advanced, symptomatic visceral spread (visceral crisis) with risk of life-threatening complications in the short term.
7. Concurrent malignancy of any site, except adequately controlled limited basal cell carcinoma or squamous-cell carcinoma of the skin, in situ melanoma or carcinoma in situ of the cervix.
8. Active cardiac disease or a history of cardiac dysfunction including any of the following:

   1. History of angina pectoris, symptomatic pericarditis, or myocardial infarction within 12 months prior to study entry
   2. History of documented congestive heart failure (New York Heart Association functional classification III-IV)
   3. Documented cardiomyopathy
   4. QTc > 480 msec as measured by Bazett's formula, family or personal history of long or short QT syndrome, Brugada syndrome or known history of QTc prolongation or Torsade de Pointes.
   5. Uncontrolled hypertension.
9. Patients being treated with drugs recognized as strong inhibitors or inducers of the isoenzyme CYP3A (including, but not limited, to - see table 6 - Rifabutin, Rifampicin, Clarithromycin, Ketoconazole, Itraconazole, Voriconazole, Ritonavir, Telithromycin) continuously for at least 7 days during any time period in the last 2 weeks prior to randomization.
10. Subjects with known dihydropyrimidine dehydrogenase (DHPD) deficiency or previous severe reactions to a fluoropyrimidine.
11. Known abnormalities in coagulation such as bleeding diathesis or ongoing treatment with anticoagulants that preclude intramuscular administration of drugs.
12. Ongoing pregnancy or lactation.
13. Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.
14. A previous metastatic tumor biopsy reported to be negative for both estrogen receptor and progesterone receptor (i.e. <1% for both), or positive for HER2 status (amplified ERBB2).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS), as assessed locally by the investigator. | Time from the date of randomization to the date of progression, assessed up to 5 years.
  Time to progression will be measured according to the RECIST criteria (version 1.1). Response criteria are essentially based on a set of measurable lesions identified at baseline as target lesions, and - together with other lesions that are denoted as non-target lesions - followed until disease progression.

SECONDARY OUTCOMES:
Health related quality of life score EuroQol (EQ-5D) | Baseline to progression up to 2 years
  Change from baseline to Health related quality of life score EuroQol (EQ-5D)
Health related quality of life score EORTC QLQ-C30 | Baseline to progression up to 2 years
  European Organisation for Research and Treatment of Cancer Quality of Life Instrument (EORTC QLQ-C30).
Health related quality of life score EORTC QLQ-BR23 | Baseline to progression up to 2 years
  European Organisation for Research and Treatment of Cancer Breast Cancer Module (EORTC QLQ-BR23).
Correlation of efficacy measures with tumor Biomarkers | Correlative analyses will be performed after the end of the trial. PFS is defined as time from the date of randomization to the date of progression assessed up to 5 years..
  PgR IHC status (10% cut-off), will be correlated with PFS
Correlation of efficacy measures with tumor Biomarkers | Correlative analyses will be performed after the end of the trial. PFS is defined as time from the date of randomization to the date of progression assessed up to 5 years.
  Ki67 IHC status, will be correlated with PFS
Correlation of efficacy measures with tumor Biomarkers | Correlative analyses will be performed after the end of the trial. PFS is defined as time from the date of randomization to the date of progression assessed up to 5 years.
  ESR1 DNA somatic mutation status, will be correlated with PFS
Correlation of efficacy measures with tumor Biomarkers | Correlative analyses will be performed after the end of the trial. PFS is defined as time from the date of randomization to the date of progression assessed up to 5 years.
  Somatic mutations in cancer genes identified by sequencing, will be correlated with PFS
Correlation of efficacy measures with tumor Biomarkers | Correlative analyses will be performed after the end of the trial. PFS is defined as time from the date of randomization to the date of progression assessed up to 5 years.
  SET index, will be correlated with PFS
Overall survival (OS) | Time from randomization to death from any cause, assessed up to 5 years.
  Overall survival from time of randomization to death from any cause.
1-year survival | Time from randomization to death from any cause, assessed up to 5 years.
  1-year survival rate from time of randomization to death from any cause.
2-year survival | Time from randomization to death from any cause, assessed up to 5 years.
  2-year survival rate from time of randomization to death from any cause.
Objective response | From randomization until end of treatment, assessed up to 5 years.
  Objective tumor response will be measured according to the RECIST criteria (version 1.1). Response criteria are essentially based on a set of measurable lesions identified at baseline as target lesions, and - together with other lesions that are denoted as non-target lesions - followed until disease progression.
Duration of response | From randomization until end of treatment, up to 5 years.
  Response duration will be measured from the time measurement criteria for complete response (CR)/ partial response (PR) (whichever is first recorded) are first met until the first date that recurrent or progressive disease is objectively documented.
Clinical Benefit Rate | From randomization until end of treatment, up to 5 years.
  Clinical Benefit Rate is defined as CR+PR+stable disease (SD) for > 24 weeks
Frequency of adverse events (AE) | From randomization until 28 days after the last dose of study medication, assessed up to 5 years.
  Adverse events will be recorded and graded according to Common Terminology Criteria for Adverse Events (CTCAE) v. 4.0

CONTACTS AND LOCATIONS:
Locations (9):
- Sweden (5):
  - Sahlgrenska University Hospital, Gothenburg
  - Skåne University Hospital, Malmo
  - S:t Görans Hospital, Stockholm
  - Karolinska University Hospital, Stockholm
  - Uppsala University Hospital, Uppsala
- United Kingdom (4):
  - NHS Grampian, Aberdeen
  - Western General Hospital, Edinburgh
  - Beatson, Glasgow
  - NHS Ayshire and Arran, Kilmarnock